CLINICAL TRIAL: NCT07301177
Title: AtMS for Alleviating Posttraumatic Peripheral Neuropathic Pain (PTP-NP)
Brief Title: DoD AtMS for Posttraumatic Peripheral Neuropathic Pain
Acronym: PTP-NP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: H240010; HT94252410300 (Other Grant/Funding Number: Department of Defense (DoD))
Record Dates: First submitted 2025-07-09; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Peripheral Neuropathic Pain; Peripheral Neuropathy; Peripheral Neuropathy Due to Surgical Trauma; Peripheral Neuropathy Due to Physical Trauma
Keywords: adaptative transcutaneous magnetic stimulation (AtMS); fixed transcutaneous magnetic stimulation (ftMS); transcutaneous magnetic stimulation (tMS); peripheral neuropathy; neuropathy; pain
MeSH Terms: conditions — Peripheral Nervous System Diseases; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Adaptive transcutaneous magnetic stimulation (AtMS) (Active Comparator): The adaptive transcutaneous magnetic stimulation (AtMS) arm uses a patient machine interface (PMI) to determine what intensity to set the study tMS treatments. Treatment is then performed with an active tMS coil.
  Interventions: Device: Transcutaneous magnetic stimulation (tMS); Device: Patient Machine Interface (PMI)
- Fixed transcutaneous magnetic stimulation (FtMS) (Active Comparator): The fixed transcutaneous magnetic stimulation (FtMS) arm uses a patient machine interface (PMI) to determine an intensity which is then multiplied by 1.5 during the first treatment session. This calculated intensity is used for every treatment session going forward, although the subject will still engage with the PMI every session. Treatments are performed using an active tMS coil.
  Interventions: Device: Transcutaneous magnetic stimulation (tMS); Device: Patient Machine Interface (PMI)
- Sham transcutaneous magnetic stimulation (Sham-tMS) (Sham Comparator): The sham transcutaneous magnetic stimulation (Sham-tMS) arm uses the patient machine interface (PMI) to determine the intensity to set the study tMS treatments for each visit. Treatment is performed using a sham tMS coil that sounds and feels the same.
  Interventions: Device: Sham transcutaneous magnetic stimulation (Sham-tMS); Device: Patient Machine Interface (PMI)

INTERVENTIONS:
Device: Transcutaneous magnetic stimulation (tMS) — Active tMS will be given at different PTP-NP sites with an active tMS coil.
  Arms: Adaptive transcutaneous magnetic stimulation (AtMS); Fixed transcutaneous magnetic stimulation (FtMS)
Device: Sham transcutaneous magnetic stimulation (Sham-tMS) — Sham-tMS will be given at different PTP-NP sites with a sham tMS coil. All parameters of the treatment will appear identical to the active treatment.
  Arms: Sham transcutaneous magnetic stimulation (Sham-tMS)
Device: Patient Machine Interface (PMI) — The PMI will be used to help determine intensities for tMS treatments.

SUMMARY:
The goal of this clinical trial is to learn if adaptative transcutaneous magnetic stimulation (AtMS) works to reduce pain caused by post-traumatic peripheral neuropathic pain (PTP-NP) within Veterans and/or active duty military personnel. It will also learn about the safety of AtMS. The main questions it aims to answer are:

1. What are the effects of adaptative tMS (AtMS) in alleviating patients' PTP-NP compared to fixed tMS (FtMS) and Sham-tMS?
2. What are the effects of AtMS in improving functions in patients suffering from PTP-NP compared to FtMS and Sham-tMS?
3. What are the effects of AtMS in improving mood in patients suffering from PTP NP compared FtMS and Sham-tMS?

Researchers will compare AtMS, FtMS and Sham-tMS to see if AtMS is the best form of tMS in treating PTP-NP.

Participants will undergo the following:

1. Receive a total of 8 AtMS, FtMS, or Sham-tMS treatments over 16 weeks.
2. Visit the clinic a total of 12 times for assessments, check ups, and treatments.
3. Keep a daily diary of their PTP-NP intensity, sleep interference, and pain medications used.

DETAILED DESCRIPTION:
This study will be enrolling a total of 144 veterans or active military over a 4 year period at the VA San Diego Healthcare System (VASDHS). Participants will be randomized into one of three groups:

Group A: AtMS Group B: FtMS Group C: Sham-tMS

Individual participation will consist of 12 visits to the VASDHS over the course of 5 months. The visits will be divided into the following phases:

1. PRE-TREATMENT ASSESSMENTS PHASE (weeks 1-2) which consists of Visit 1 (Screening Visit) and Visit 2 (Baseline Assessments)
2. INDUCTION TREATMENT PHASE (weeks 3-4) consists of Visits 3-7 (5 weekday tMS sessions at >24 and <72 hours apart); and
3. POST-TREATMENT ASSESSMENTS AND MAINTENANCE TREATMENT PHASE (weeks 6-20) consists of 2 initial biweekly post-induction treatment assessments and maintenance treatments (Visits 8 and 9), and two additional monthly post-induction treatment assessments and maintenance treatments (Visits 10 and 11) and one final study visit (Visit 12)

ELIGIBILITY:
Inclusion Criteria:

* Veterans (men or women) of any race or ethnicity who are at least 18 years of age
* Chronic peripheral neuropathic pain present for more than 4 months after a traumatic or surgical event per medical history
* Have an average daily Numerical Pain Rating Scale (NPRS) score > 3
* At least one negative or positive sensory sign or symptom confined to innervation territory of the lesioned nervous structure
* Prior diagnostic tests confirming lesion or disease explaining neuropathic

Exclusion Criteria:

* Pregnancy
* Subjects with central neuropathic pain (ex: due to diabetic peripheral neuropathy, HIV, chemo/anti-viral therapy, carpal tunnel syndrome, post-traumatic pain classified as central rather than peripheral)
* Subjects with pain due to Complex Regional Pain Syndrome
* Phantom limb pain after amputation (stump pain and phantom sensation are allowed)
* Subjects with skin conditions in the affected dermatome
* Subjects with other pain such as lumbar or cervical radiculopathy that may confound assessment
* Any subject considered at risk of suicide
* Use of prohibited medications in the absence of appropriate washout periods
* Participation in any other clinical trial within the 30 days prior to screening and/or during participation in this study
* Heart pacemaker
* Subjects with a current diagnosis of DSM-IV-TR Axis I disorder (GAD & MDD are allowed if clinically stable)
* Subjects with pending lawsuits related to injury
* Subjects who have previously received either transcranial or transcutaneous magnetic stimulation therapy in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Neuropathic Pain Rating | From enrollment to the end of treatment at 20 weeks
  0 is equivalent to no neuropathic pain and 10 indicates the worst possible neuropathic pain
Mood | From baseline to the end of treatment at 20 weeks
  Hamilton Rating Scale for Depression (HRSD) an interviewed asks 21 questions about mood, sleep, appetite, and other symptoms related to depression. The interviewer rates the severity of each symptom based on a pre-defined scale of 0-4. The scores for each item are then summed to produce a total score.
  The total score on the HAM-D is used to assess the severity of depression. Lower scores indicate less severe depression, while higher scores indicate more severe depression.
  Typical scoring interpretations: Below 7: Absence or remission of depression; 7-17: Mild depression; 18-24: Moderate depression; 25 and above: Severe depression
Quality of Life (Sleep Interference) | From enrollment to the end of treatment at 20 weeks
  Daily Sleep Interference Log measures how much neuropathic pain impacts the patients sleep each night. The log is ranked on a 0 to 10 scale, 0 being pain didn't interfere with sleep and 10 being pain completely interfered with sleep, with a lower score representing a better outcome.
Functionality - Absenteeism | From baseline to the end of treatment at 20 weeks
  Work Productivity and Activity Impairment Questionnaire (WPAI-SHP version 2) metric 1:
  Absenteeism (the percentage of work time missed);
  ***Only those being employed provided answer for absenteeism***
  WPAI absenteeism scores are based 2-items (2 and 4); a score cannot be calculated if there is a missing response to the corresponding item. Question 2 represents time in hours lost due to health reasons while question 4 represents the time spent working. Time lost is divided by the total time (sum of 2 and 4) and then multiplied by 100 to express as a percentage.
  All WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity
Functionality - Presenteeism | From baseline to the end of treatment at 20 weeks
  Work Productivity and Activity Impairment Questionnaire (WPAI-SHP version 2) metric 2:
  Presenteeism (the percentage of impairment experienced while at work);
  ***Only those being employed provided answer for presenteeism***
  WPAI presenteeism scores are based on 1-item (5) which is divided by 10 and later multiplied by 100 to express as a percentage; a score cannot be calculated if there is a missing response to the corresponding item.
  WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity
Functionality - Overall work Productivity Impairment | From baseline to the end of treatment at 20 weeks
  Work Productivity and Activity Impairment Questionnaire (WPAI-SHP version 2) metric 3:
  Overall work productivity loss (an estimate of combination of absenteeism and presenteeism);
  ***Only those being employed provided answer for absenteeism {Q2/(Q2+Q4)}, presenteeism {Q5/10}***
  WPAI overall work productivity scores are computed based on absenteeism and presenteeism scores, using the following formula, Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4)))x(Q5/10)], and then being multiplied by 100 to express as a percentage; a score cannot be calculated if there is a missing response to the corresponding item.
  WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity
Functionality - Activity Impairment | From baseline to the end of treatment at 20 weeks
  Work Productivity and Activity Impairment Questionnaire (WPAI-SHP version 2) metric 4:
  Activity impairment (the percentage of impairment in daily activities)
  ***Only those being employed provided answer for absenteeism, presenteeism, and overall work impairment***
  WPAI activity impairment scores are based on 1-item (item 6) which is divided by 10 and later multiplied by 100 to express as a percentage; a score cannot be calculated if there is a missing response to the corresponding item.
  WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity

SECONDARY OUTCOMES:
Neuropathic Pain Medication Usage | From enrollment to the end of treatment at 20 weeks
  Neuropathic Pain Medication Logs will measure changes in daily neuropathic pain. The log will record if daily neuropathic pain medications are used, the medication name(s), the strength(s) measured in mg, quantity measured by number of pills/sprays/etc. As well as if additional non-daily, typically OTC, pain medications were taken for neuropathy, the medication name(s), strength(s) measured in mg, quantity measured by number of pills/spray/etc.
  For this outcome, increases in any medication as well as new medications will be marked as "more" and numerically described with 1; decreases will be marked as "less" and numerically described as -1; no change will result in a 0. Total change will be summed per visit and later used as a percentage of participants positive (representing an increase in medication us) or negative (decrease in medication use) change.
  Any negative score will be considered a favorable outcome.
Allodynia Area Mapping (Von Frey) | From baseline to the end of treatment at 20 weeks
  von Frey 5.18 monofilament will be used to measure/map (cm²) out an area of neuropathic allodynia. The instrument will be used by pressing them against the neuropathic pain area and marking roughly 8 points with each. Then the points will be traced on two separate translucent papers, one for each instrument, to create two rough shapes to measure the areas. The area of the shape will be measured using a Compensating Polar Planimeter.
Allodynia Area Mapping (paint brush) | From baseline to the end of treatment at 20 weeks
  Paintbrush will be used to measure/map (cm²) out an area of neuropathic allodynia. The instrument will be used by pressing them against the neuropathic pain area and marking roughly 8 points with each. Then the points will be traced on two separate translucent papers, one for each instrument, to create two rough shapes to measure the areas. The area of the shapes will be measured using a Compensating Polar Planimeter.
QST Temperature Thresholds | From baseline to end of treatment at 20 weeks
  Thermal Sensory Analyzer (Medoc Advanced Medical Systems, Minneapolis) will be used to measure cool, warm, cold, and hot temperature (°C) thresholds.
  The participant will first be asked to press the button when the increasing hot temperature becomes uncomfortable. This will be done 3 times and averaged to establish a threshold for the next portion.
  The thermode will heat up to the threshold temperature and remain their for a period of time. The participant will then rate their pain experienced via MVAS scale (0-10) with a 0 describing no pain and a 10 describing the worst pain experienced.
  A lower pain score will represent a better outcome and a higher score will represent a worse outcome.
von Frey Monofilament Threshold | From baseline to end of the treatment at 20 weeks
  Different sized von Frey monofilament (e.g, 5.18) will be used to determine the participants physical pain sensation threshold to the von Frey monofilaments. The von Frey monofilaments will pressed against the neuropathic pain area one by one from smallest to largest until the participants expresses they can feel a sensation of physical pain in the neuropathic area caused by the von Frey monofilament.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Y Leung, M.D., Principal Investigator — Veterans Medical Research Foundation (VMRF)
Locations (1):
- Veterans Medical Center - San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No